CLINICAL TRIAL: NCT00325377
Title: A Randomized Sham-Controlled Clinical Study to Evaluate the Effects of the Magnetic Molecular Energizer (MME)on Chronic Low Back Pain
Brief Title: The Effects of the MME Procedure on Chronic Low Back Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Advanced Magnetic Research Institute International (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMRI-LBP-002
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain; pain; magnetism; electromagnetic fields; visual analogue pain scale
MeSH Terms: conditions — Low Back Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: MME Procedure

SUMMARY:
The purpose of this study is to test whether or not the Magnetic Molecular Energizer (MME) device provides a well tolerated and effective intervention to reduce pain, pain-related symptoms and improve ability to function in those diagnosed with the condition "Chronic Low Back Pain" (chronic LBP).

DETAILED DESCRIPTION:
Pilot studies conducted by AMRI International suggest that 0.5T static magnetic field energy as supplied by the investigational device Magnetic Molecular Energizer (MME) may be effective for relieving chronic low back pain that has been persistent despite conventional therapy. This study is is a randomized, sham-controlled trial intended to show whether or not the MME intervention is an effective, well tolerated intervention for the reduction of pain, pain related symptoms and improved ability to function in those diagnosed with the condition, chronic low back pain.

The MME procedure consists of laying on a treatment bed with the individual's body positioned between two large, electromagnetic coils that create a very strong (0.3T - 0.5T) magnetic field that passes through the body. The device bears a superficial resemblance to an open MRI machine. The field is focused on the low back area. The total intervention time for the study is 140 hr of MME exposure, consisting of 8 - 12 hrs per day for 12 - 18 consecutive days or nights. Participants with be assessed prior to starting the intervention by history and physical exam conducted by one of the physician investigators, assessing pain level by using a visual analogue pain scale, assessing functional ability using the Oswestry Low Back Pain Disability Index questionnaire and assessment of cutaneous perception threshold (CPT) using the Neurometer device.

Pain scale levels will be assessed daily throughout the intervention period. At the conclusion of the intervention period, CPT testing will be repeated. One month after the intervention, the Oswestry Low Back Pain Disability Index questionnaire will be mailed to the participant. The final evaluation will be six months after the intervention. The participant is to return to the clinic and repeat CPT testing, report pain levels and complete the Oswestry Low Back Pain Disability Index questionnaire.

The targeted enrollment for the trial is 100 participants. The participants will be randomized so that 50 receive the active procedure and 50 will receive a sham procedure. The sham procedure is provided by a MME device that has been disabled so that the machine appears to turn on, but no magnetic field is produced. When the final post-intervention follow-up has been completed the participants will be informed whether they received the active or sham procedure. Those who received the sham procedure will be offered to receive the active procedure if they desire. The same evaluations will be repeated with this cross-over group, but the data will be reported separately from the main trial results.

Participants are not asked to discontinue their usual medications or treatments for their low back pain. Medication usage will be assessed to see if there is any change in usage pattern associated with the procedure.

ELIGIBILITY:
Inclusion Criteria:

* daily low back pain of at least 3 months duration
* stable neurologic status
* prior medical work up and trial of standard medical therapy

Exclusion Criteria:

* progressive neurologic deficits
* neurologic deficits in the legs due to a medical condition other than the back
* severe obesity (BMI > 34.9)
* long acting narcotics
* severe spinal stenosis (fixed obstruction of the spinal canal)
* pacemakers, defibrillators, implanted medication pump, spinal cord stimulator or shrapnel
* low back screws, rods, artificial discs or cages
* fibromyalgia
* pregnancy
* an open insurance claim or pending legal claim or settlement related to the back pain, or retired on back-related disability, or receiving disability pension related to the back problem

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-04; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
reduction in pain
improved ability to function

SECONDARY OUTCOMES:
tolerability to procedure
neurologic stability
reduction in pain medication

CONTACTS AND LOCATIONS:
Overall Officials: Wayne R Bonlie, M.D., Study Director — AMRI International; Dean R Bonlie, DDS, Study Chair — AMRI International
Locations (5):
- United States (5):
  - AMRI Arizona, Tucson, Arizona
  - AMRI Michegan, Sterling Heights, Michigan
  - AMRI North Carolina, Mocksville, North Carolina
  - AMRI NW Ohio, Toledo, Ohio
  - AMRI WA, Renton, Washington